CLINICAL TRIAL: NCT04710004
Title: Electrophysiological Biomarkers During Invasive Monitoring of Mesial Temporal Lobe Epilepsy Patients.
Brief Title: Electrophysiological Biomarkers in MTLE Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to secure effort for testing.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Robert Gross, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001554
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Mesial Temporal Lobe Epilepsy
Keywords: Epilepsy; Biomarkers
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Brain stimulation via clinically implanted electrodes (Experimental): Brain will be stimulated in different patterns including synchronized or asynchronous current.
  Interventions: Device: Asynchronous distributed multi-electrode stimulation (ADMES) using an implantable neurostimulation device

INTERVENTIONS:
Device: Asynchronous distributed multi-electrode stimulation (ADMES) using an implantable neurostimulation device — Participants will receive asynchronous pulses distributed across a multi-electrode array of 16 micro-electrodes and stimulating at low (theta) frequencies.
  Other Names: ADMES

SUMMARY:
The investigators plan to enroll individuals with medical temporal lobe epilepsy who are undergoing surgical workup with clinically implanted intracranial electrodes. The study intends to administer computerized memory tasks and stimulation during the intracranial Electroencephalography (EEG) monitoring period.

DETAILED DESCRIPTION:
This is a nonrandomized interventional trial that will apply brain stimulation via clinically implanted intracranial electrodes to subjects with medial temporal lobe epilepsy with the purpose of identifying biomarkers related to the pre-ictal state; to perform an acute parameter search to determine the stimulation pattern that most effectively modifies these biomarkers and to identify changes in memory (free recall) during asynchronous distributed multi-electrode stimulation (ADMES).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male or female, aged 18-65
3. Diagnosed with lesional or non-lesional mesial temporal (hippocampal) seizure onset confirmed on SEEG monitoring
4. Implanted with depth electrodes for localization of seizure onset with multiple hippocampal electrode arrays

Exclusion criteria:

1. Any patient who is unwilling or unable to provide consent
2. Women who are pregnant
3. Patients under 18 years
4. Incarcerated persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gross, MD, Principal Investigator — Emory University
Locations (1):
- Epilepsy monitoring unit (EMU) at Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brain Stimulation Via Clinically Implanted Electrodes
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brain Stimulation Via Clinically Implanted Electrodes
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Intracranial EEG Recording: Spectral Power From Baseline
Description: Spectral power will be compared between baseline/sham and stimulation trials to determine if asynchronous stimulation modulates spectral power during the preictal, ictal or post ictal states. Spectral power is measured in microvolts. A change in either direction from baseline is associated with a better outcome.
Time Frame: Baseline, up to 6 weeks postintervention
Population: No data collected. Subject was discharged before testing could be completed.
Arm/Group | Brain Stimulation Via Clinically Implanted Electrodes
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Intracranial EEG Recording: Synchrony From Baseline
Description: Synchrony will be compared between baseline/sham and stimulation trials to determine if asynchronous stimulation modulates synchrony during the preictal, ictal or post ictal states. Synchrony is a measure of how any pair of regions communicate with one another. Synchrony is measured as the correlation [-1 to 1] between two time series.
  The investigators anticipate that a decrease in synchrony (correlation approaching 0) is associated with improved outcome.
Time Frame: Baseline, up to 6 weeks postintervention
Population: No data collected. Subject was discharged before testing could be completed.
Arm/Group | Brain Stimulation Via Clinically Implanted Electrodes
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Memory During Brain Stimulation From Baseline
Description: Patients will be asked to recall a list of words after a 20-second delay in which they will do simple math problems to ensure long-term memory encoding. Three ~1-2-hour sessions will be performed; each session will consist of 24 free recall tasks (12 during ADMES and 12 with no stimulation). The memory score will be assessed as the percentage correct out of 12. The higher the percentage recalled, the better the score.
Time Frame: Baseline, up to 6 weeks postintervention
Population: No data collected. Subject was discharged before testing could be completed.
Arm/Group | Brain Stimulation Via Clinically Implanted Electrodes
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 16 days
Arm/Group | Brain Stimulation Via Clinically Implanted Electrodes
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT04710004/Prot_SAP_000.pdf